CLINICAL TRIAL: NCT02191774
Title: Medical Abortion up to 10 Weeks Gestation at Home
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lena Marions, Associate professor, senior consultant, Karolinska Institutet
Other Study IDs: Marions 2014 1.2; 2013-004749-18 (EudraCT Number)
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy Complications; Legally Induced Abortion Without Mention of Complication
Keywords: Medical abortion; Home abortion
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gestational length up to 63 days: Medical abortion at home using 200 mg of Mifepristone orally at the clinic followed by 0.8 mg Cytotec vaginally at home 48 hours later
  Interventions: Procedure: Medical abortion at home
- Gestational length 64-70 days: Medical abortion at home using 200 mg of Mifepristone orally at the clinic followed by 0.8 mg Cytotec vaginally at home 48 hours later
  Interventions: Procedure: Medical abortion at home

INTERVENTIONS:
Procedure: Medical abortion at home — Medical abortion using Mifepristone at the clinic followed by Cytotec at home

SUMMARY:
Medical abortion performed in the womens home has shown to be safe and acceptable up to 9 weeks of gestation. Our project is aiming to confirm our hypothesis that it is equally effective, safe and acceptable when the gestation is more advanced, up to 10 weeks of gestation.

DETAILED DESCRIPTION:
The study will include 600 women opting for medical abortion. Women wanting to perform the last part of the abortion in their homes will be invited to participate. 300 women with a pregnancy up to 9 weeks of gestation (63 days) will be compared to 300 women with a gestation length between 64 and 70 days of gestation. The primary endpoints will be number of patients with an incomplete abortion, with a need for surgical or pharmaceutical intervention.

Secondary endpoints include duration of bleeding, acceptance and satisfaction with the method and number of additional visits to the clinic/facility.

The study will be performed in five abortion clinics in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Requesting and eligible for medical abortion
* Confirmed intrauterine pregnancy
* Gestational length no more than 70 days
* Hemoglobin over 100g/l

Exclusion Criteria:

* Anemia
* Contraindication to mifepristone (steroid-dependant cancer, porphyria)
* Breast feeding
* Advanced pregnancy (>70 days)
* Known liver disease
* Bleeding disorder
* Arterial hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with an unwanted pregnancy opting for medical abortion
Sampling Method: Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Number of incomplete abortions | 4 weeks after treatment
  Need for surgical or pharmaceutical intervention

SECONDARY OUTCOMES:
Duration of bleeding | 4 weeks after treatment
  Measured by diary and questionnaires
Acceptance and satisfaction of treatment | 4 weeks after treatment
  Questionnaires
Number of additional visits to the clinic | 4 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lena Marions, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Podolskyi V, Gemzell-Danielsson K, Maltzman LL, Marions L. Effectiveness and acceptability of home use of misoprostol for medical abortion up to 10 weeks of pregnancy. Acta Obstet Gynecol Scand. 2023 May;102(5):541-548. doi: 10.1111/aogs.14549. Epub 2023 Mar 18. PMID 36933004